CLINICAL TRIAL: NCT04280042
Title: Long-term Outcomes in Long Standing Persistent Atrial Fibrillation Following Catheter Or Thoracoscopic Surgical Ablation : Extended Follow-Up Of CASA-AF Randomised Controlled Trial
Brief Title: Long-term Outcomes in Long Standing Persistent Atrial Fibrillation
Acronym: LoTO_CASA_AF
Status: Completed | Type: Observational
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other); Brighton and Sussex University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 271930
Record Dates: First submitted 2020-02-18; First posted 2020-02-21 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Long Standing Persistent Atrial Fibrillation
Keywords: atrial fibrillation; thoracoscopic surgical AF ablation; catheter ablation; implanted loop recorder
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Serum samples to assess the values of a range of biomarkers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Thoracoscopic surgical ablation: Participants in CASA AF Trial who underwent thoracoscopic surgical ablation to treat their long standing persistent AF will be asked to continue downloading the data from their implanted loop recorder, attend two hospital appointments (at 24 and 36 months post ablation) to complete questionnaires, have an ECG, a blood test and report current medications they use.
- Cather ablation: Participants in CASA AF Trial who underwent conventional catheter ablation to treat their long standing persistent AF will be asked to continue downloading the data from their implanted loop recorder, attend two hospital appointments (at 24 and 36 months post ablation) to complete questionnaires, have an ECG, a blood test and report current medications they use.

SUMMARY:
Atrial fibrillation (AF) is a condition detected as an irregular heartbeat. It is the most common rhythm disturbance worldwide which can lead to significant symptoms and serious health problems (stroke and heart failure). The longer a person has AF, the more difficult it is to restore a normal heart rhythm. Those with continuous AF for longer than a year are described as having longstanding persistent AF (LSPAF). This is the most challenging type of AF to treat and medications are often not effective. Apart from medications patients with LSPAF may be offered a medical procedure to help improve their symptoms. It involves putting a flexible thin tube (catheter) into a blood vessel in the groin and up into the heart to destroy the tissue causing irregular heart beat. This procedure has modest success in improving symptoms in the long term. Recently, keyhole surgery has been used for these patients and evidence shows that it is better than the catheter procedure. However, we do not know how well people are doing beyond one year. Feedback from a patient focus group suggested that knowing the long-term results of these two procedures is important to help them make an informed choice when it comes to treatment. In this study we propose to continue monitoring patients from a randomised clinical trial (CASA AF RCT) who have already had one of the procedures. They have a small heartbeat monitor implanted under the skin with a battery life of around 3 years. We will be able to look at their heart rhythm data for the duration of this period and detect the return of the fibrillation if it happens.

DETAILED DESCRIPTION:
This study involves participants from the randomised clinical trial which was just completed (CASA AF RCT: NCT02755688; ISRCTN18250790 ). They have undergone relevant ablation procedures in a randomised fashion and completed 12 months follow up. At the last study visit they signed a consent form to confirm that they have agreed to keep implanted loop recorder for the duration of its battery life time (approximately 3 years). They have also continued to regularly transfer data from their implanted loop recorder to the secure server where it is regularly reviewed. This group of patients is now a unique cohort whose follow up data is invaluable for additional research. For this study we will ask for their written consent and apart from analysing their heart rhythm data we will arrange two hospital visits with some additional tests and completion of questionnaires.

The principal objective of the study is to compare the long-term effectiveness of thoracoscopic surgical ablation and percutaneous catheter ablation, the two procedures available for treatment of atrial fibrillation in patients with longstanding persistent AF (LSPAF). There is some evidence that thoracoscopic surgical ablation may be better than catheter ablation in keeping the patients in regular heart rhythm after a single procedure without use of antiarrhythmic drugs in short term. In this study we plan to monitor patients who have undergone these procedures for 3 years.

Our secondary objectives are focussing on patients who had more than one procedure and/or may be using medications in order to maintain regular heart rhythm during 36 months follow up.

We will therefore look at:

1. the effectiveness of a single procedure (catheter or surgical) in maintaining normal rhythm with use of antiarrhythmic drugs.
2. the effectiveness of multiple ablative procedures in maintaining sinus rhythm with and without use of antiarrhythmic drugs.
3. the proportion of patients who are still in AF but the time they spend in it is reduced by ≥75%.

   We will also want to examine:
4. patient reported change in quality of life from baseline to 24 and 36 months after ablative treatment.
5. changes in levels of serum biomarkers from baseline to 36 months and how they relate to the freedom of arrhythmia
6. health and social care resource use and associated costs from baseline to 36 months
7. the cost-effectiveness of thoracoscopic surgical ablation compared with catheter ablation and update the health economic model developed for the main study (CASA AF RCT).

Our sample size calculations show that with an expected rate of attrition of around 20% we need 94-100 study participants to show the difference in the effectiveness of the two procedure with power of 80%, p= 0.05.

Patients participating in this extended follow-up study will attend two hospital appointments to coincide with 24 and 36 months post-ablation (± 6 months). These two visits will consist of:

1. clinical examination
2. review of concurrent medications and comorbidities
3. electrocardiogram (12 lead ECG )
4. blood test for routine biochemistry and collection of a sample for biomarkers analyses
5. completion of questionnaires to assess patients' quality of life: atrial fibrillation effect on quality of life (AFEQT), EuroQol (EQ5D5L) European Heart Rhythm Association score of atrial fibrillation (EHRA),
6. Health economic questionnaire to capture repeat procedures (ablation, direct current cardioversion and AF-related emergency care)

For the duration of the extended follow-up, once a week patients will download data from their implantable loop recorders which have algorithms that are specific for atrial arrhythmias (atrial fibrillation, atrial tachycardia, atrial flutter). Patients remotely download their data to the Medtronic (MyCarelinkTM) secure server. These data will be reviewed centrally every month by a dedicated Research Fellow. Patients will be contacted monthly by telephone to ensure compliance and to discuss any rhythm abnormalities detected in these data that require review of treatment/ management. Patients will be able to contact the research team if they experience symptoms of atrial arrhythmias. The implanted loop recorder data can be interrogated remotely, and appropriate advice regarding treatment given based on data review.

ELIGIBILITY:
Inclusion Criteria:

CASA-AF RCT participants who have undergone ablative procedure to treat their LSPAF, completed 12 months follow up and consented to keep their implanted loop recorders in situ with weekly data downloads.

Exclusion Criteria:

There are no exclusion criteria for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with long standing persistent atrial fibrillation who took part in the CASA AF clinical trial and underwent one of the intervetions: catheter ablation or surgical thoracoscopic ablation. These patients have agreed to keep their implanted loop recorders and continued to dowload their data.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Effectiveness of a single ablative procedure | over the duration of the followup period (24 months)
  Freedom from continuous atrial arrhythmia (≥120 seconds in duration) recorded by implantable loop recorder or other clinically indicated rhythm recording device and absence of anti-arrhythmic drugs on concurrent medications form.

SECONDARY OUTCOMES:
Reduction of burden of atrial fibrillation | over the duration of the followup period (24 months)
  Proportion of patients who experience recurrence of atrial arrhythmias but are in sinus rhythm 75% of the time or more
AF related quality of life | at 24 and 36 months from the ablative treatment
  Measurement of changes in overall AFEQT scores (18 questions) and treatment satisfaction scores (2 questions) from baseline to two follow up time points
Quality of life assessment | at 24 and 36 months from the ablative treatment
  EQ5D5L questionnaires (descriptive and analogue scale) will be completed at baseline and two follow up timepoints. Changes in scores on both scales will be used to assess and quantify patients' health outcome
Changes in concentration of serum biomarkers (pg/ml) | from baseline to 36 months after the ablative procedure
  Serum assays for different biomarkers (pg/ml) will be performed at baseline and compared to the concentrations in samples collected at follow up visits. Increase (or decrease) of the biomarkers' concentration will be related to freedom from arrhythmia during follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Tom Wong, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton and Harefield NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No